CLINICAL TRIAL: NCT05271370
Title: An Extension Protocol for Virologically Suppressed Subjects Who Successfully Completed PRO140_CD03 Study
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: FDA required the sponsor to halt enrollment in the trial and transition participants to available therapies for the treatment of their disease. The trial was subsequently terminated once participants were transitioned.
Sponsor: CytoDyn, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO 140_CD03 Extension
Record Dates: First submitted 2022-01-13; First posted 2022-03-09 (Actual); Results first posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — leronlimab

STUDY DESIGN:
Intervention Model Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- PRO 140 350 mg (Experimental): PRO 140 350mg weekly SC injection.
  Interventions: Drug: PRO 140 350
- PRO 140 525 mg (Experimental): PRO 140 525mg weekly SC injection.
  Interventions: Drug: PRO 140 525
- PRO 140 700 mg (Experimental): PRO 140 700mg weekly SC injection.
  Interventions: Drug: PRO 140 700

INTERVENTIONS:
Drug: PRO 140 350 — Pro140 SC injection 350 mg
  Other Names: leronlimab
  Arms: PRO 140 350 mg
Drug: PRO 140 525 — 525 mg
  Other Names: leronlimab
  Arms: PRO 140 525 mg
Drug: PRO 140 700 — 700 mg
  Other Names: leronlimab
  Arms: PRO 140 700 mg

SUMMARY:
This study is a Phase 2b/3 multi-center extension study designed to evaluate the long term antiviral activity, safety, and tolerability of the strategy of continuing PRO 140 350mg, 525mg, or 700mg SC (subcutaneous) monotherapy to maintain viral suppression after initial 48 weeks in virologically suppressed subjects.

Consenting subjects will continue weekly PRO 140 350mg, 525mg, or 700mg monotherapy during the Treatment Extension Phase with the one-week overlap of existing retroviral regimen and PRO 140 350mg, 525mg, or 700 mg at the end of the treatment in subjects who do not experience virologic failure.

DETAILED DESCRIPTION:
The objective is to assess the long-term safety of using PRO 140 350mg, 525mg, or 700mg SC as single-agent maintenance therapy for the chronic suppression of CCR5-tropic HIV-1 infection.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have completed 48 weeks of treatment in PRO140_CD03 study.
2. Last known Plasma HIV-1 RNA < 50 copies/mL within PRO140_CD03 study.
3. Both male and female patients and their partners of childbearing potential must agree to use 2 medically accepted methods of contraception (e.g., barrier contraceptives [male condom, female condom, or diaphragm with a spermicidal gel], hormonal contraceptives [implants, injectables, combination oral contraceptives, transdermal patches, or contraceptive rings], and intrauterine devices) during the course of the study (excluding women who are not of childbearing potential and men who have been sterilized). Females of childbearing potential must have a negative serum pregnancy test at Screening visit and negative urine pregnancy test prior to receiving the first dose of study drug.
4. Willing and able to participate in all aspects of the study, including use of SC medication, completion of subjective evaluations, attendance at scheduled clinic visits, and compliance with all protocol requirements as evidenced by providing written informed consent.

Exclusion Criteria:

1. Not currently enrolled in PRO140_CD03 study.
2. Any active infection or malignancy requiring acute therapy (with the exception of local cutaneous Kaposi's sarcoma).
3. Females who are pregnant, lactating, or breastfeeding, or who plan to become pregnant during the study.
4. Subjects weighing < 35kg.
5. History of anaphylaxis to any oral or parenteral drugs.
6. History of Bleeding Disorder or patients on anti-coagulant therapy (except aspirin).

   Note: Subjects with well-controlled bleeding disorder while on stable anti-coagulant therapy dose with documented stable INRs can be enrolled as per discretion of the Investigator.
7. Any other clinical condition that, in the Investigator's judgment, would potentially compromise study compliance or the ability to evaluate safety/efficacy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Lalezari, MD, Principal Investigator — CytoDyn, Inc.
Locations (1):
- Quest Clinical Research, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- PRO 140 350 mg: PRO 140 350mg weekly SQ injection.
  PRO 140 350: Pro140 SC injection 350 mg
- PRO 140 525 mg: PRO 140 525mg weekly SQ injection.
  PRO 140 525: 525 mg
- PRO 140 700 mg: PRO 140 700mg weekly SQ injection.
  PRO 140 700: 700 mg
Period: Overall Study
Arm/Group | PRO 140 350 mg | PRO 140 525 mg | PRO 140 700 mg
Started | 8 | 18 | 30
Completed | 0 | 2 | 1
Not Completed | 8 | 16 | 29
Not completed — Study early termination | 8 | 16 | 29

BASELINE CHARACTERISTICS:
Population: All patients who received at least one dose of PRO 140 (leronlimab) were included in the baseline analysis population. Study was early terminated.
Groups:
- Total: Total of all reporting groups
Arm/Group | PRO 140 350 mg | PRO 140 525 mg | PRO 140 700 mg | Total
Number analyzed (Participants) | 8 | 18 | 30 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 17 | 28 | 52
  >=65 years | 1 | 1 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.88 (8.37) | 47.17 (11.94) | 47.77 (13.10) | 49.30 (12.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 0 | 4
  Male | 7 | 15 | 30 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 4 | 5 | 9
  Not Hispanic or Latino | 8 | 14 | 25 | 47
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 4 | 7
  White | 7 | 13 | 26 | 46
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 18 | 30 | 56

OUTCOME MEASURES:

1. Primary Outcome: Long Term Clinical Safety of PRO 140 Monotherapy by Assessing the Number of Participants With Grade 2, 3 or 4 Adverse Events as Defined by the DAIDS Adverse Event Scale, and the Number of Participants With Treatment-emergent Serious Adverse Events.
Description: The Division of AIDS (DAIDS) grading table provides an adverse event severity grading scale ranging from grades 1 to 5 with descriptions for each adverse event based on the following general guidelines:
  * Grade 1 indicates a mild event
  * Grade 2 indicates a moderate event
  * Grade 3 indicates a severe event
  * Grade 4 indicates a potentially life-threatening event
  * Grade 5 indicates death (Note: This grade is not specifically listed on each page of the grading table). Treatment-Emergent Serious Adverse Events (TESAEs) are defined as serious adverse events with an onset on or after the first treatment.
Time Frame: From TE1 (first treatment administration) to last treatment visit, up to 197 weeks
Population: The safety population is defined as all subjects who received at least one dose of PRO 140 within the PRO 140_CD03 extension study.
Measure: Number; unit: participants
Arm/Group | PRO 140 350 mg | PRO 140 525 mg | PRO 140 700 mg
Number analyzed (Participants) | 8 | 18 | 30
participants
  Participants with Grade 2, 3, or 4 AEs | 5 | 6 | 6
  Participants with TESAEs | 3 | 5 | 2

2. Primary Outcome: Proportion of Participants Experiencing Virologic Failure for All Subjects Within Each Treatment Group.
Description: Virological failure is defined as two consecutive HIV-1 RNA levels of ≥ 200 copies/mL for all subjects and within each treatment group.
Time Frame: From TE1 (first treatment administration) to last treatment visit, up to 197 weeks
Population: The analysis population is defined as all subjects who enrolled in the study and received at least one dose of PRO 140.
Measure: Number; unit: proportion of participants
Arm/Group | PRO 140 350 mg | PRO 140 525 mg | PRO 140 700 mg
Number analyzed (Participants) | 8 | 18 | 30
proportion of participants | 0 | 0.17 | 0.37

3. Secondary Outcome: Time to Virologic Failure After Initiating PRO 140 Monotherapy for All Subjects Within Each Treatment Group.
Description: Virological failure (VF) is defined as two consecutive HIV-1 RNA levels of ≥ 200 copies/mL for all subjects and within each treatment group. The date of VF event is defined as the date of the second assessment of the two (2) consecutive HIV-1 RNA levels of >= 200 copies/mL when virological failure is confirmed. Subjects who did not have VF, the last visit date will be used as the date of the event.
Time Frame: From TE1 (first treatment administration) to last treatment visit, up to 197 weeks
Population: The analysis population is defined as all subjects who enrolled in the study and received at least one dose of PRO 140.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | PRO 140 350 mg | PRO 140 525 mg | PRO 140 700 mg
Number analyzed (Participants) | 8 | 18 | 30
days | 1148.88 (457.15) | 735.67 (326.71) | 582.00 (407.71)

4. Secondary Outcome: Proportion of Participants Achieving Viral Re-suppression After Experiencing Virologic Failure Within Each Treatment Group.
Description: Viral re-suppression is defined as having HIV-1 RNA levels of < 50 copies/mL after experiencing virologic failure within each treatment group.
Time Frame: From TE1 (first treatment administration) to last treatment visit, up to 197 weeks
Population: The population includes all subjects who experienced virologic failure for each treatment group. No virologic failure was reported in the 350 mg treatment group.
Measure: Number; unit: Portion of Participants
Arm/Group | PRO 140 350 mg | PRO 140 525 mg | PRO 140 700 mg
Number analyzed (Participants) | 0 | 3 | 11
Portion of Participants |  | 1 | 0.9

5. Secondary Outcome: Time to Achieving Viral Re-suppression After Experiencing Virologic Failure Within Each Treatment Group.
Description: as for outcome 4
Time Frame: From TE1 (first treatment administration) to last treatment visit, up to 197 weeks
Population: The population includes all subjects who experienced virologic failure and re-suppression for each treatment group. No virologic failure was reported in the 350 mg treatment group.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | PRO 140 350 mg | PRO 140 525 mg | PRO 140 700 mg
Number analyzed (Participants) | 0 | 3 | 10
days |  | 100.33 (33.48) | 136.71 (127.68)

6. Secondary Outcome: Proportion of Virologic Failure Subjects Achieving Viral Re-suppression With Re-initiation of Previous Baseline Antiretroviral Regimen Within Each Treatment Group.
Description: Viral re-suppression is defined as having HIV-1 RNA levels of < 50 copies/mL after experiencing virologic failure within each treatment group. Subjects who experienced virologic failure during the treatment phase had an option to re-initiate their PRO 140 regimen to their previous baseline or dose escalate to the next dose level.
Time Frame: From TE1 (first treatment administration) to last treatment visit, up to 197 weeks
Population: The population includes all subjects who experienced virologic failure and achieved viral re-suppression for each treatment group. No virologic failure was reported in the 350 mg treatment group.
Measure: Number; unit: proportion of participants
Arm/Group | PRO 140 350 mg | PRO 140 525 mg | PRO 140 700 mg
Number analyzed (Participants) | 0 | 3 | 10
proportion of participants |  | 0.33 | 0.78

7. Secondary Outcome: Mean Change in CD4 Cell Count, at Each Visit Within the Treatment Phase for All Subjects Within Each Treatment Group
Description: The change from baseline in CD4 cell count was summarized for each visit during the treatment phase for each treatment group. The time-weighted mean of change of the post baseline (visit TE1) values was calculated. The time-weighted mean was adjusted AUC (area under the curve) by time.
Time Frame: From TE1 (first treatment administration) to last treatment visit, up to 197 weeks
Population: The analysis population is defined as all subjects who enrolled in the study and received at least one dose of PRO 140. Subjects who had undefined change from baseline due to missing data were excluded from the analysis population.
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | PRO 140 350 mg | PRO 140 525 mg | PRO 140 700 mg
Number analyzed (Participants) | 8 | 18 | 27
cells/uL | 0.62 (2.60) | -0.14 (2.59) | 0.58 (2.32)

ADVERSE EVENTS:
Time Frame: Report initiation for all adverse events began at the time of the first treatment extension visit and continued up until the final study visit (up to approximately 197 weeks).
Description: AEs were elicited through direct questioning and subject reports. Any abnormalities in visit evaluations, physical examination findings or laboratory results that the Investigator believed clinically significant to the research subject and that occurred after initiation of the first study treatment were reported as AEs.
Arm/Group | PRO 140 350 mg | PRO 140 525 mg | PRO 140 700 mg
All-Cause Mortality (participants affected / at risk) | 1/8 | 1/18 | 0/30
Serious Adverse Events (participants affected / at risk) | 3/8 | 5/18 | 2/30
Other Adverse Events (participants affected / at risk) | 6/8 | 9/18 | 18/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRO 140 350 mg (N=8) | PRO 140 525 mg (N=18) | PRO 140 700 mg (N=30)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lacunar infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
Pancreatitis necrotising (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Polymyositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRO 140 350 mg (N=8) | PRO 140 525 mg (N=18) | PRO 140 700 mg (N=30)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 2 (5) | 0 (0) | 0 (0)
Anal chlamydia infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (8) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Chlamydial infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Cluster headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Colonoscopy (Investigations) | 1 (1) | 0 (0) | 0 (0)
Computerised tomogram abdomen (Investigations) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (3) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 2 (4) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 2 (2) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Ear Discomfort (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Ear Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (6) | 0 (0)
Endoscopy (Investigations) | 1 (1) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Essential tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (3) | 1 (1) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Heat exhaustion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (2) | 3 (3)
Injection site haematoma (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Menopause (Social circumstances) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Mitral valve Prolapse (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Mucous stools (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (5) | 3 (5) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1)
Ocular hypertension (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oliguria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Onychomycosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Oropharyngeal gonococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (3) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Polycythaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Retching (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 3 (4) | 1 (1) | 0 (0)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Skin bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (4) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Syphilis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 4 (7) | 5 (7)
Urethritis chlamydial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urine flow decreased (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
FDA required the sponsor to halt enrollment in the trial and transition participants to available therapies for the treatment of their disease. The trial was subsequently terminated once participants were transitioned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-30): https://cdn.clinicaltrials.gov/large-docs/70/NCT05271370/Prot_SAP_000.pdf